CLINICAL TRIAL: NCT04579120
Title: Neuroimaging in Healthy Aging and Senile Dementia (HASD_IND)
Acronym: HASD_PIB_IND
Status: Recruiting | Type: Observational
Sponsor: Tammie L. S. Benzinger, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Tammie L. S. Benzinger, MD, PhD, Professor of Radiology & Neurological Surgery, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: 201906009
Record Dates: First submitted 2020-08-12; First posted 2020-10-08 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
Keywords: Dementia; Neuro-Degenerative Disease; Amyloid Plaque; Mild Cognitive Impairment; Brain Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia; Plaque, Amyloid; Cognitive Dysfunction; Brain Diseases | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole; 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- African American: African American participants receiving [11C]-Pittsburgh Compound B ([11C]PiB) F 18 AV-1451 (Flortaucipir) for imaging.
  Interventions: Drug: [11C]-Pittsburgh Compound B ([11C]PiB); Drug: F 18 AV-1451 (Flortaucipir)
- Non-Hispanic White: Non-Hispanic White participants receiving [11C]-Pittsburgh Compound B ([11C]PiB) F 18 AV-1451 (Flortaucipir) for imaging.
  Interventions: Drug: [11C]-Pittsburgh Compound B ([11C]PiB); Drug: F 18 AV-1451 (Flortaucipir)

INTERVENTIONS:
Drug: [11C]-Pittsburgh Compound B ([11C]PiB) — A dosage range between 6.0 - 20.0 mCi (222-740 MBq) is planned for [11C] PIB. A PET-certified medical professional will prepare and administer the [11C] PIB tracer. Prior to the administration, the dosage will be assayed in a dose calibrator and diluted with 0.9% sodium chloride (normal saline) up to a total 20 mL syringe volume. Participants will receive a maximum intravenous bolus injection of 20.0 mCi of [11C] PIB followed by a 10 mL 0.9% sodium chloride (normal saline) flush.
  Other Names: PiB
Drug: F 18 AV-1451 (Flortaucipir) — A dosage range between 6.5 - 10.0 mCi (240-370MBq) is planned for [18F] AV-1451. A PET-certified medical professional will prepare and administer the [18F] AV-1451tracer. Prior to the administration, the dosage will be assayed in a dose calibrator. The volume of 18F-AV-1451 dose should not be adjusted by adding normal saline to the syringe. Participants will receive a maximum intravenous bolus injection of 10.0 mCi of [18F] AV-1451 followed by a 10 mL flush of 0.9% sodium chloride (normal saline).
  Other Names: F 18 AV-1451

SUMMARY:
To identify factors that signal the transition from asymptomatic (preclinical) to symptomatic Alzheimer disease (AD).

DETAILED DESCRIPTION:
The purpose of this research study is to evaluate the structure and function of the brain in healthy aging and early Alzheimer's disease using positron emission tomography (PET), magnetic resonance imaging (MRI), and computed tomography (CT) imaging. The study involves imaging the brain to detect the presence of amyloid deposits (plaques in the brain). Amyloid is a protein that may be related to dementia of Alzheimer's disease (DAT).

This study will use radioactive tracers called C-11 Pittsburgh Compound B (PIB) and F 18/ AV-1451 (Flortaucipir) which binds to beta amyloid and tau in the brain. These compounds are considered investigational, which means that they have not been approved by the United States Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, any race
* Age > 18 years
* Participation in one of the ongoing projects affiliated with the Knight ADRC at Washington University and referred by the MAP staff and a Washington University physician.
* Normal cognition or early-stage symptomatic AD
* Willing and able to undergo study procedures.
* Capacity to give informed consent and follow study procedures

Exclusion Criteria:

* Has any condition that, in the Investigator's opinion, could increase risk to the participant, limit the participant's ability to tolerate the research procedures, or interfere with the collection/analysis of the data (e.g., participants with severe chronic back pain might not be able to lie still during the scanning procedures);
* Has hypersensitivity to either AV-1451 or PIB or any of its excipients;
* Contraindications to PET, CT or MRI (e.g. electronic medical devices, inability to lie still for extended periods) that make it unsafe for the individual to participate;
* Severe claustrophobia;
* Currently pregnant or breast-feeding. Women must agree to avoid becoming pregnant and must agree to refrain from sexual activity or to use reliable contraceptive methods for 24 hours following administration of Flortaucipir injection;
* Must not have participated in any clinical trial involving a study drug or device within the 30-days prior to study enrollment;
* Must not participate in another drug or device study prior to the end of this study participation;
* Current or recent (within 12 months prior to screening) participation in research studies involving radioactive agents such that the total research-related radiation dose to the participant in any given year would exceed the limits set forth in the U.S. Code of Federal Regulations (CFR) Title 21 Section 361.1.

https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/CFRSearch.cfm?FR=361.1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are referred from the Washington University Knight Alzheimer's Disease Research Center (ADRC). The ADRC is responsible for the recruitment, enrollment, and maintenance of the Total Registry (TR). The Knight ADRC primarily recruits participants by means of word of mouth and public service announcements from the greater metropolitan St. Louis area. A small percentage (~17%) of participants are referred by a Washington University physician.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
AD Biomarkers seen on Amyloid PET at Baseline and Years 1, 2, and/or 3 | 5 years
  This Project aims to identify factors that signal the transition from asymptomatic (preclinical) to symptomatic Alzheimer disease (AD). This will be done by comparing imaging biomarkers seen with amyloid PET and the tracer C-11 PIB at baseline to imaging biomarkers collected longitudinally, at years 1, 2, and/or 3.
AD Biomarkers seen on Tau PET at Baseline and Years 1, 2, and/or 3 | 5 years
  This Project aims to identify factors that signal the transition from asymptomatic (preclinical) to symptomatic Alzheimer disease (AD). This will be done by comparing imaging biomarkers seen with tau PET and the tracer Flortaucipir at baseline to imaging biomarkers collected longitudinally, at years 1, 2, and/or 3.
AD Biomarkers seen on MRI at Baseline and Years 1, 2, and/or 3 | 5 years
  This Project aims to identify factors that signal the transition from asymptomatic (preclinical) to symptomatic Alzheimer disease (AD). This will be done by comparing imaging biomarkers seen with MRI at baseline to imaging biomarkers collected longitudinally, at years 1, 2, and/or 3.
Compare and Correlate Predictive Ability of Biomarkers Seen with Different Imaging Variables for Onset of Symptoms | 5 years
  This project aims to compare and correlate the predictive ability of baseline values and rates of change of molecular biomarkers of AD for onset of AD symptoms with other variables. Variables obtained in this project include: 1) volumetric MRI, 2) MRI measures of vascular burden, 3) functional MRI, 4) amyloid PET, and 5) tau PET.

SECONDARY OUTCOMES:
Compare and Correlate Predictive Ability of Biomarkers Seen with Other Types of Variables for Onset of Symptoms | 5 years
  This project aims to compare and correlate the predictive ability of baseline values and rates of change of molecular biomarkers of AD for onset of AD symptoms with other variables obtained through Knight ADRC data sharing, which include, 1) clinical (demographic information, socioeconomic status, Clinical Dementia Rating, etiology of cognitive disorder (when present), and comorbid disorders, including cardiovascular disease); 2) cross-sectional and longitudinal cognitive performance, 3) indicators of sleep disruption 4) APOE genotype and genetic variants associated with resilience novel CSF analytes of neurofilament light chain, neurogranin, and SNAP-25 as markers of axonal and synaptic injury.
Disparities for molecular biomarkers of AD in non-Hispanic white (NHW) and African American (AA) older adults | 5 years
  The study will also focus on disparities for molecular biomarkers of AD in non-Hispanic white (NHW) and African American (AA) older adults. Aim 2 will compare the risk (or the hazard) of developing AD symptoms by race, and will treat death as a potential competing risk in the progression of dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Benzinger, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
We will share imaging data with other researchers. They may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at Washington University, at other research centers and institutions, or industry sponsors of research. We may also share research data with large data repositories (a repository is a database of information) for broad sharing with the research community. If individual research data is placed in one of these repositories only qualified researchers, who have received prior approval from individuals that monitor the use of the data, will be able to look at your information. The shared information will not include names but may be linked by a global unique identifier (GUID) number.